CLINICAL TRIAL: NCT06356285
Title: How Can we Frame Antimicrobial Resistance in the Best Way to Inspire Behaviour Change? An Online Randomised Controlled Trial.
Brief Title: Testing New Ways to Name Antimicrobial Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: The Behavioural Insights Team (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 6995049
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Antimicrobial Resistance; Attitude to Health
Keywords: Antimicrobial Resistance; Behaviour Change

STUDY DESIGN:
Intervention Model Description: This study has been designed as a four-armed online randomised control trial (RCT). This will be conducted using Predictiv, an online platform for running behavioural experiments built by the Behavioural Insights Team The 4,000 participants will be randomised in a 1:1:1:1 ratio to one of four trial arms.
Who Masked: Participant
Masking Description: Participants will be blinded to the study arm that they have been assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Arm - Antimicrobial Resistance (No Intervention): Participants will be shown an image of a poster at a bus stop. This will contain information about antibiotics, and will have the words "Antimicrobial Resistance" at the top.
- Intervention Arm 1 - Superbugs (Experimental): Participants will be shown an image of a poster at a bus stop. This will contain information about antibiotics, and will have the word "Superbugs" at the top.
  Interventions: Behavioral: Presentation of Antimicrobial Resistance
- Intervention Arm 2 - Antibiotic Resistance (Experimental): Participants will be shown an image of a poster at a bus stop. This will contain information about antibiotics, and will have the words "Antibiotic Resistance" at the top.
  Interventions: Behavioral: Presentation of Antimicrobial Resistance
- Intervention Arm 3 - Antibiotic Crisis (Experimental): Participants will be shown an image of a poster at a bus stop. This will contain information about antibiotics, and will have the words "The Antibiotic Crisis" at the top.
  Interventions: Behavioral: Presentation of Antimicrobial Resistance

INTERVENTIONS:
Behavioral: Presentation of Antimicrobial Resistance — Participants will be presented with a poster containing information about antibiotics, each intervention poster will have a different name at the top, representing a new way to frame antimicrobial resistance.
  Arms: Intervention Arm 1 - Superbugs; Intervention Arm 2 - Antibiotic Resistance; Intervention Arm 3 - Antibiotic Crisis

SUMMARY:
This study aims to investigate the public's views on antibiotics and the impact of different ways to name the potential consequences of antibiotics not working in the future. It is known that current ways to name this don't resonate well with the public, and the study team have worked with members of the public through focus groups and community workshops to develop new ways of describing this in a process of co-design. This study aims to test four different ways of presenting this potential crisis to the public, some of which are new communication strategies designed by the public themselves, to evaluate which are the most memorable and investigate the impact on behaviour change.

Adults aged over 18, living in the United Kingdom, who have already signed up to a market panel research company will be eligible to participate in this study.

Participants will be invited to complete a short online survey (this should take around five minutes), advertised to them by the market research panel they have already signed up to. This survey is completely anonymous, and contains some multiple-choice questions, and some that require a short free text response. At the start of the survey one of the four ways to name AMR will be presented to participants in the form of a poster.

This study aims to result in an improved understanding regarding the general public's understanding of antibiotic use and investigate the impact of communication on behaviour change. The data from this study may be used to inform future public health campaigns on this topic and improve the use of antibiotics.

This study will be conducted online using the Predictiv platform, an online platform built by the Behavioural Insights Team. The study is being run in collaboration between the Behavioural Insights Team and the Institute of Global Health Innovation at Imperial College London.

Is it anticipated that the survey will open in April 2024 and be open until recruitment of 4000 participants is complete. This is expected to take 4-6 weeks.

DETAILED DESCRIPTION:
Antimicrobial resistance (AMR) refers to the process by which bacteria become resistant to antibiotics, rendering them ineffective in treating infections. Public behaviour change is needed to use antibiotics more sparingly and wisely (for example, only taking them when needed and finishing the course). However, studies and public engagement work have shown that the current language around the crisis of AMR is not well known or understood by the general public. It is felt to be too scientific, not memorable, and doesn't convey sufficient meaning to inspire behaviour change.

Building on previous studies, this project aims to identify whether different ways to present or frame Antimicrobial Resistance (AMR) can lead to improved comprehension and change attitudes towards the crisis. Through extensive public engagement and involvement work three different ways to frame AMR to the public have been developed. One of these ways is a novel name developed through co-design with public members, and the other two were existing terms that the public believed were better than AMR during our engagement activities.

An online randomised controlled trial (RCT) has been designed to test these three names against the control of AMR/Antimicrobial resistance, to see if they can improve comprehension, attitudes towards and recall of the subject.

This online RCT will be delivered in collaboration with the Behavioural Insights Team using their well established online platform, called Predictiv. 4,000 participants will be recruited (to be representative of the UK population). They will see one of our four names (this will be presented in the typical community setting of seeing a poster at a bus stop), and be asked to complete a short five minute survey, answering a series of questions to explore their understanding of the topic and their future attitudes to antibiotic use.

Statistical analysis will be conducted to see which of the four communication strategies were most effective across the different outcomes, helping us to understand which communication strategies for AMR are most useful at inspiring behaviour change. Data will additionally be analysed to explore whether different messaging strategies are more effective in certain population subgroups - for example by age or previous antibiotic use.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged over 18
* Resident in the United Kingdom (UK)
* Have passed the attention check at the start of the online survey.

Exclusion Criteria:

* Individuals not signed up a market research panel, and will therefore not have access to the online survey
* Those resident outside the UK
* Those who fail the attention check at the start of the online survey.
* Individuals aged under 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4296 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate Grailey, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No personal IPD will be collected in this study. Aggregate participant data will be shared between the Behavioural Insights Team and Imperial College London

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Arm - Antimicrobial Resistance | Intervention Arm 1 - Superbugs | Intervention Arm 2 - Antibiotic Resistance | Intervention Arm 3 - Antibiotic Crisis
Started | 1055 | 1113 | 1092 | 1036
Completed | 1055 | 1113 | 1092 | 1036
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adults residing in the United Kingdom who accessed the online survey and passed the attention check.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm - Antimicrobial Resistance | Intervention Arm 1 - Superbugs | Intervention Arm 2 - Antibiotic Resistance | Intervention Arm 3 - Antibiotic Crisis | Total
Number analyzed (Participants) | 1055 | 1113 | 1092 | 1036 | 4296
Age, Customized [Count of Participants; unit: Participants]
  18-24 | 121 | 129 | 114 | 123 | 487
  25-39 | 279 | 281 | 272 | 258 | 1090
  40-54 | 283 | 304 | 295 | 296 | 1178
  55+ | 372 | 399 | 411 | 359 | 1541
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 565 | 580 | 541 | 538 | 2224
  Female | 487 | 526 | 543 | 494 | 2050
  Other | 3 | 7 | 8 | 4 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 93 | 98 | 75 | 84 | 350
  Black | 31 | 31 | 39 | 24 | 125
  Mixed / Other | 39 | 55 | 38 | 45 | 177
  White | 892 | 929 | 940 | 883 | 3644
Region of Enrollment [Number; unit: participants]
  United Kingdom | 1055 | 1113 | 1092 | 1036 | 4296

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Correct Answers by Participants on Questions Designed to Evaluate Attitudes Towards Antimicrobial Resistance (Sentiment)
Description: Evaluation of participant's attitudes towards antimicrobial resistance, related to questions within the survey that assess sentiment (including agreement that antimicrobial resistance is an urgent issue that needs to be addressed, antimicrobial resistance poses a risk to human health and antimicrobial resistance is an issue that may impact the participants own health).
  This was conducted using a quasi-binominal regression model using the sum of binary ratings of sub-sentiment questions as the primary outcome analysis.
Time Frame: 6 weeks
Population: All adults (over the age of 18, representative of the UK population) who responded to the survey question.
Measure: Number; unit: percentage of correct answers
Units Other Than Participants: Survey Answers (One per participant)
Arm/Group | Control Arm - Antimicrobial Resistance | Intervention Arm 1 - Superbugs | Intervention Arm 2 - Antibiotic Resistance | Intervention Arm 3 - Antibiotic Crisis
Number analyzed (Participants) | 1055 | 1113 | 1092 | 1036
Number analyzed (Survey Answers (One per participant)) | 1055 | 1113 | 1092 | 1036
percentage of correct answers | 81 | 83.2 | 86.3 | 85.2
Statistical Analysis 1: Comparison: Intervention Arm 1 - Superbugs vs Intervention Arm 2 - Antibiotic Resistance vs Intervention Arm 3 - Antibiotic Crisis; Test type: Equivalence — Quasibinominal models were used as the outcomes are bounded count variables. Accepting a two-sided p-value adjusted for 3 comparisons, the study was designed with 80% power to detect a minimal detectable effect size between the trial arms and control for the primary outcome; p = 0.017, Quasibinominal regression — A two-sided p-value, as shown in the table, which was adjusted for 3 comparisons; Odds Ratio, log = 0.05

2. Secondary Outcome: Percentage of Correct Answers by Participants on Questions Designed to Evaluate Comprehension of Antimicrobial Resistance
Description: Comprehension of the meaning of Antimicrobial Resistance, related to questions within the survey that evaluate comprehension (what has caused antimicrobial resistance, what is the solution to antimicrobial resistance, what antimicrobial resistance is).
  This was conducted using a quasi-binominal regression model using the number of correct answers to comprehension questions.
Time Frame: 6 weeks
Population: Adults residing in the UK aged over 18, passed attention check
Measure: Number; unit: Percentage of correct answers
Units Other Than Participants: Survey Answers (one per participant)
Arm/Group | Control Arm - Antimicrobial Resistance | Intervention Arm 1 - Superbugs | Intervention Arm 2 - Antibiotic Resistance | Intervention Arm 3 - Antibiotic Crisis
Number analyzed (Participants) | 1055 | 1113 | 1092 | 1036
Number analyzed (Survey Answers (one per participant)) | 1055 | 1113 | 1092 | 1036
Percentage of correct answers | 63.3 | 65.1 | 66.0 | 65.4

3. Secondary Outcome: Percentage of Participants Who Stated They Would Request Antibiotics
Description: Intention regarding antibiotic use in the context of antimicrobial resistance related to questions within the survey that evaluate intent - asking participants about whether they would request antibiotics in certain scenarios.
  This was conducted using a separate logistic regression for each scenario (binary - Yes or No).
Time Frame: 6 weeks
Population: Adults residing in the UK aged over 18, passed attention check
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Survey Answers (One per participant)
Arm/Group | Control Arm - Antimicrobial Resistance | Intervention Arm 1 - Superbugs | Intervention Arm 2 - Antibiotic Resistance | Intervention Arm 3 - Antibiotic Crisis
Number analyzed (Participants) | 1055 | 1113 | 1092 | 1036
Number analyzed (Survey Answers (One per participant)) | 1055 | 1113 | 1092 | 1036
Percentage of participants | 8.7 | 8.5 | 8.8 | 8.4

4. Secondary Outcome: Percentage of Participants Who Correctly Recalled the Terminology Related to Antimicrobial Resistance
Description: Recall of the term used to describe antimicrobial resistance in the intervention. This was conducted using a separate logistic regression for each question (asking about recall of the name at the top of the poster and the content of the poster) (binary - Yes or No).
Time Frame: 6 weeks
Population: Adults residing in the UK aged over 18, passed attention check
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Survey Answers (One per participant)
Arm/Group | Control Arm - Antimicrobial Resistance | Intervention Arm 1 - Superbugs | Intervention Arm 2 - Antibiotic Resistance | Intervention Arm 3 - Antibiotic Crisis
Number analyzed (Participants) | 1055 | 1113 | 1092 | 1036
Number analyzed (Survey Answers (One per participant)) | 1055 | 1113 | 1092 | 1036
Percentage of participants | 72 | 65.4 | 79 | 74.5

ADVERSE EVENTS:
Time Frame: Serious and other [non-serious] adverse events were not collected or assessed as part of the study: No adverse event data were collected. Given this is an online survey, with no personal identifying information gathered the risk of serious adverse events or all-cause mortality is zero.
Description: Given this is an online survey, with no personal identifying information gathered the risk of serious adverse events or all-cause mortality is zero
Groups:
- Control Arm - Antimicrobial Resistance; Intervention Arm 1 - Superbugs; Intervention Arm 2 - Antibiotic Resistance; Intervention Arm 3 - Antibiotic Crisis: Serious and other [non-serious] adverse events were not collected or assessed as part of the study
Arm/Group | Control Arm - Antimicrobial Resistance | Intervention Arm 1 - Superbugs | Intervention Arm 2 - Antibiotic Resistance | Intervention Arm 3 - Antibiotic Crisis
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT06356285/Prot_SAP_000.pdf